CLINICAL TRIAL: NCT05048524
Title: Peri-operative S-1/Leucovorin, Oxaliplatin and Gemcitabine (SLOG) for Localized Pancreatic Cancer
Brief Title: Peri-operative SLOG for Localized Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Responsible Party: Principal Investigator, Yung-Yeh Su, Principal investigator, National Health Research Institutes, Taiwan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLOG
Record Dates: First submitted 2021-08-30; First posted 2021-09-17 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Pancreas Cancer
Keywords: Neoadjuvant Therapy; SLOG; S-1; Leucovorin; Oxaliplatin; Gemcitabine
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — S 1 (combination); Leucovorin; Oxaliplatin; Gemcitabine

STUDY DESIGN:
Intervention Model Description: Two cohorts: unresectable and resectable
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SLOG (Experimental)
  Interventions: Drug: S-1, leucovorin, oxaliplatin and gemcitabine

INTERVENTIONS:
Drug: S-1, leucovorin, oxaliplatin and gemcitabine — Gemcitabine 800 mg/m2 on day 1, oxaliplatin 85 mg/m2 on day 1, S-1 orally 80-120 mg/day [depending on patient's body surface area (BSA)] on day 1 to 7 and leucovorin 30mg BID day 1 to 7 on in a 2-week cycle. The dose of S-1 is defined as follows:
  * BSA < 1.25 m2: 80 mg/day
  * 1.25 m2 ≤ BSA < 1.5 m2: 100 mg/day
  * BSA ≥ 1.5 m2: 120 mg/day

SUMMARY:
1. To evaluate the efficacy of neoadjuvant chemotherapy SLOG in localized pancreatic cancer
2. To evaluate the safety profile in patients with pancreatic cancer who receive neoadjuvant SLOG
3. To collect tumor tissue and peripheral blood samples from the patients for a comprehensive biomarker evaluation

DETAILED DESCRIPTION:
The role of neoadjuvant treatment in pancreatic adenocarcinoma is still under debate due to a relative lack of robust data compared with other gastrointestinal cancers. According to 2020 NCCN guidelines, neoadjuvant is now the accepted approach for borderline resectable (BR) disease, while upfront surgery is still the recommendation for resectable disease except in cases with high risk features. Another important advantage of treatment with neoadjuvant treatment is an increase in the proportion of patients who receive chemotherapy. Traditionally, only patients with a good performance status and a good recovery after surgery are treated with adjuvant chemotherapy. About 45% of patients do not receive adjuvant chemotherapy after resection due to poor performance status, postoperative morbidity, or early progression of disease. A small cohort study using total neoadjuvant FOLFIRINOX for borderline resectable pancreatic cancer yielded a promising result but the tolerability of FOLFIRINOX limited the use of this regimen in Asian population. In previous T1211 clinical trial, the SLOG regimen showed comparable efficacy with a better safety profile in metastatic pancreatic cancer. This phase II trial will evaluate the feasibility of SLOG regimen in patients with localized pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

A. Localized resectable or potentially resectable pancreatic cancer as determined by image modality; resectability is determined by the treating surgeon No prior treatment for pancreatic cancer

B. Patients must agree to receive biopsy for histological diagnosis and provide residual tissue for biomarker analysis before chemotherapy

C. Patients must agree to provide tissue for biomarker analysis after neoadjuvant chemotherapy, either surgical specimen or follow-up biopsy in unsectable disease

D. At least one measurable lesion according to RECIST version 1.1

E. Ability to understand and willingness to sign a written informed consent document.

F. Eastern Cooperative Oncology Group (ECOG) performance status 0-1

G. Age of 20 years or above

H. Life expectancy of at least 12 weeks

I. Adequate organ function as defined by the following criteria:

* absolute neutrophil count (ANC) ≥ 1,500/mm3
* hemoglobin level ≥ 9 g/dL
* platelet count ≥ 100,000/mm3
* total bilirubin < 2 mg/dL
* aspartate aminotransferase (AST) / alanine aminotransferase (ALT) ≤ 3 x upper limit of normal (ULN)
* creatinine clearance rate (CCr) ≥ 50 mL/min (24-hour urine collection or calculated by Cockroft-Gault formula; male: [(140 - age) × weight (kg)]/[72 × serum creatinine(mg/dL)];female=male x 0.85

J. Patients with childbearing potential shall have effective contraception for both the patient and his or her partner during the study.

Exclusion Criteria:

A. Other malignancy within the past 5 years except for adequately treated localized skin cancer or cervical cancer in situ;

B. Presence of distant metastasis;

C. Presence of mental disease or psychotic manifestation;

D. Active or uncontrolled infection;

E. Significant medical conditions that is contraindicated to study medication or render patient at high risk from treatment complications at physician discretion

F. Pregnant women or nursing mothers, or positive pregnancy test for women of childbearing potential.

G. History of active autoimmune disease within 3 years or use of steroid more than prednisolone 10mg/day.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-09-03 (Actual); Primary Completion 2024-08-24 (Estimated); Study Completion 2025-08-24 (Estimated)

PRIMARY OUTCOMES:
The percentage of subjects with R0 resection after surgery | 1 year

SECONDARY OUTCOMES:
The percentage of subjects successfully underwent surgery after study drug treatment | 1 year
The percentage of subjects with tumor shrinkage >30% | 1 year
  according to RECIST 1.1
The percentage of subjects without tumor progression | 1 year
  tumor progression is defined as increase of size by >20% according to RECIST 1.1
Progression-free survival (PFS) of patient received study treatment | 1 year
Overall survival (OS) of patient received study treatment | 2 years
Duration of response (DOR) of patient received study treatment | 1 year
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 2 years
Biomarkers of treatment response by single cell RNA sequencing and whole exome sequencing | 4 years
  Biomarkers including but not limited to tumor mutation burden, change of immune cell proportion and percentage of T-reg in the tumor microenvironment.

CONTACTS AND LOCATIONS:
Locations (3):
- Taiwan (3):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - National Cheng-Kung University Hospital, Tainan
  - National Institute of Cancer Research, Tainan

IPD SHARING:
Plan to Share IPD: Undecided